CLINICAL TRIAL: NCT04569175
Title: Non Enhanced Labyrinth Imaging for the Detection of Endolymphatic Hydrops in Meniere's Disease "NELI Study"
Acronym: NELI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2020/25
Record Dates: First submitted 2020-09-10; First posted 2020-09-29 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Meniere Disease
Keywords: Meniere's disease; NE 3D FLAIR sequence
MeSH Terms: conditions — Meniere Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D Flair sequence (Experimental): Optimized 3D FLAIR sequence before and 4 hours after the usual care MRI (with contrast product)
  Interventions: Other: 3D Flair sequence

INTERVENTIONS:
Other: 3D Flair sequence — Optimized 3D FLAIR sequence before and 4 hours after the usual care MRI (with contrast product). All patients will have the same intervention as each patient is its own control

SUMMARY:
This study includes 30 patients with Meniere's disease confirmed with AAO-HNS criteria.

The aim of this study is to compare the new optimized 3D FLAIR sequence developed at our site with a standard 3D FLAIR sequence performed 4h after a single intravenous dose of macrocyclic gadolinium-based contrast agents for the detection of endolymphatic hydrops.

The patients will be explored with the new 3D FLAIR optimized sequence before injection (method to validate) and again 4 hours after contrast media administration with the same sequence 3D FLAIR

DETAILED DESCRIPTION:
Meniere's disease (MD) is a pathology of the inner ear defined by episodes of spontaneous vertigo usually accompanied by tinnitus, pressure within the ear and fluctuating sensorineural hearing loss.

Endolymphatic hydrops (EH) is the main pathophysiological substratum of Meniere's disease. Temporal bone MRI has long been used performed to exclude other pathologies mimicking MD, such as vestibular schwannoma or endolymphatic sac tumor.

Currently, delayed 3D-FLAIR sequence is the imaging technique of choice for the diagnosis of endolymphatic hydrops. The endolymphatic space could be assessed on MRI with 3D-FLAIR sequences delayed acquisition after the intravenous administration of gadolinium.

The saccule appears to be the most involved structure in MD. The reproducibility of the hydrops protocols with various MRI scan manufacturers is debatable.

Because endo and peri lymphatic spaces have different biochemical compositions, a new FLAIR 3D sequence on healthy volunteers can be tuned in order to separate endo and peri lymphatic spaces. The hypothesis of the study is that this new method could detect saccular hydrops with the same performances as the standard FLAIR that is done after gadolinium injection.

This study will prospectively include 30 patients with MD confirmed with AAO-HNS criteria . All patients will sign an informed consent. They will be explored with the new 3D FLAIR optimized sequence without injection (method to validate). Then, they will be injected, and they will be explored again 4 hours after contrast product administration with the same sequence (the reference method),to take advantage of the intravenous injection of gadolinium that will be performed in the care. The optimized non enhanced 3D FLAIR sequence will be compared with the reference method and with the same sequence four hours after gadolinium injection.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman
* older than 18 years old.
* Uni- or bilateral definite or probable clinical diagnosis of MD based on the AAO-HNS guidelines revised in 2015.
* Patient eligible for having contrast-enhanced MRI.
* Patient affiliated of beneficiary of health insurance
* Patient has signed the Informed consent form.

Non inclusion criteria:

* History of other pathology of the inner ear.
* History of surgery on the middle or inner ear (tympanoplasty, endolymphatic sac drainage, vestibular schwannoma).
* Pregnant (contraceptive method, HAS criteria) or nursing mothers
* Contraindications to performing MRI (pace maker, metallic shards, claustrophobia)
* Contraindications (relative) to injecting gadolinium (severe renal failure due to the risk of systemic nephrogenic fibrosis, history of allergic reaction)
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Kappa coeficient | 1 hour before baseline (usual care MRI)
  the non-inferiority of the non-enhanced Flair sequence compared to the reference technique by indirect comparison with the reference method (Kappa coefficient > or equal to 0.81).

SECONDARY OUTCOMES:
inter-observer correlation | 1 hour before baseline, baseline, 4 hours after baseline
  inter-observer correlation coefficient (weighted Kappa).

OTHER OUTCOMES:
Meniere disease categorization | 1 hour before baseline, baseline, 4 hours after baseline
  Patient's clinical categorization according to the diagnostic criteria for Meniere's disease formulated by the Classification Committee of the Barany Society in 2015 : definite Meniere's disease and probable Meniere's disease.
Degree of endolymphatic hydrops | 1 hour before baseline, baseline, 4 hours after baseline
  degree of endolymphatic hydrops: grade I/II/III
Volume of endolymphatic hydrops | 1 hour before baseline, baseline, 4 hours after baseline
  Volume of endolymphatic hydrops: quantification (mm3)
Peak width | 1 hour before baseline, baseline, 4 hours after baseline
  peak width in multifrequency tympanometry: average +/- standard deviation
Resonant frequency | 1 hour before baseline, baseline, 4 hours after baseline
  Resonant frequency: 0 to 2000 Hz

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No